CLINICAL TRIAL: NCT03840226
Title: The Impact of Magnesium Oxide Monohydrate Compared to Placebo on Exercise Tolerance, Quality of Life and Clinical Outcomes in Chronic Heart Failure Patients
Brief Title: The Impact of Magnesium on Exercise Tolerance, Quality of Life and Clinical Outcomes in Chronic Heart Failure Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Naveh Pharma (1996) Ltd. (Unknown)
Responsible Party: Principal Investigator, Michael Shechter, Director, Clinical Research Unit, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHEBA-18-5464-MS-CTIL
Record Dates: First submitted 2019-02-09; First posted 2019-02-15 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Magnesium Deficiency; Heart Failure
Keywords: magnesium; heart failure
MeSH Terms: conditions — Magnesium Deficiency; Heart Failure | interventions — Magnesium Oxide

STUDY DESIGN:
Intervention Model Description: The aim of the study is to test The impact of magnum versus placebo, on six-minute and clinical outcomes of patients with CHF (level 2-4).
  The Primary endpoints are:
  1. Improvement in Six-Minute walk test.
  2. Improvement in clinical outcomes: death, CHF hospitalization, revascularization etc.
  To test the hypothesis that the six-minute results between the two study groups are different, with significance level of 5% and power of at least 80%, we use the t-test. Based on Monica et al (2001), the mean six-minute results among these patients is 218 with SD=28. for an expected difference of at least 10 meter, we need a sample size of 125 patients in each group.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium (Active Comparator): oral magnesium oxide tablets [Magnox 520 TM (magnesium oxide monohydrate, 520 mg/day of elemental magnesium), Naveh Pharma, Israel]
  Interventions: Drug: Magnesium Oxide
- Placebo (Placebo Comparator): Placebo tablets
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Placebo Oral Tablet — Placebo tablets
  Other Names: Placebo
  Arms: Placebo
Drug: Magnesium Oxide — Magnesium tablets
  Other Names: Magnox 520 TM
  Arms: Magnesium

SUMMARY:
Magnesium supplementation could improve cardiac performance. Patients with chronic heart failure (CHF) are magnesium deficient and we hypothesized that 1 year supplementation of oral magnesium comparted to placebo will improve exercise duration time and quality of life.

DETAILED DESCRIPTION:
Magnesium supplementation improves myocardial metabolism, inhibits calcium accumulation and myocardial cell death; it improves vascular tone, peripheral vascular resistance, afterload and cardiac output, reduces cardiac arrhythmias and improves lipid metabolism. Magnesium also reduces vulnerability to oxygen-derived free radicals, improves human endothelial function and inhibits platelet function. Patients with chronic heart failure (CHF) are magnesium deficient. The activation of the renin-angiotensin-aldosterone system and the use of diuretics are associated with depletion of potassium and magnesium in CHF. Magnesium deficiency stimulates aldosterone production and secretion, while magnesium infusion decreases aldosterone production production by inhibiting cellular calcium influx. Adamopoulos et al recently found that CHF in patients [mainly New York Heart Association (NYHA) II-II] with low serum magnesium ≤ 2 mEq/L was associated with increased cardiovascular mortality (but had no association with cardiovascular hospitalization) compared to those with serum magnesium > 2 mEq/L in a long-term follow-up of 36 months, suggesting that most of these deaths were likely sudden (arrhythmic) in nature.

Furthermore, Stepura and Martynow demonstrated that oral magnesium orotate used as adjuvant therapy in severe NYHA IV CHF patients increased 1-year survival rate and improved clinical symptoms and patient's quality of life compared to placebo. The investigators hypothesized that 1-year supplementation of oral magnesium compared to placebo to CHF patients will improve exercise duration time and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* CHF patients NYHA II-IV > 3 months
* Diuretic therapy > 3 months
* Signed informed consent

Exclusion Criteria:

* chronic renal failure (serum creatinine > 3 mg/dL)
* AMI/ACS< 3 months from randomization
* Cardiac or other organ transplantation
* Uncontrolled hypo/hyperthyroidism
* Chronic diarrhea
* Life expectancy < 1 year
* Known psychiatric disease which inhibits patient's enrollment to the study
* Inability to come for follow-up visits
* Any planned operation/invasive procedures in the near 6 months
* Uncontrolled cardiac arrhythmias
* Inability to perform 6 minute walk testing
* Any participation in another interventional clinical trial < 1 month from randomization
* Any malignancy with life expectancy < 1 year Any AV Block> 2 degree without a pacemaker

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2019-08-25 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in exercise duration time | 1 year
  Improvement in 6-minute walking testing (any improvemnt of length in meters from baseline). The outcome will be measured in meters and the higher is better from baseline. A 10% higher distance from baseline will be considered significant improvement.
Qaulity of life | 1 year
  Improvement in quality of life by Minisota living with Heart Failure Questionnaire. The scale is in points and the higher scale the better. Any improvement in at least 10% from baseline will be considered a significant improvement.

SECONDARY OUTCOMES:
Improvment in the number of hospitalizations for heart failure | 1 year
  All hospitalizations for worsening of heart failure will be counted and recorded and the number of hospitalizations for heart failure will be conted in the magnesium compared to the placebo arms.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Shechter, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Leviev Heart Center, Chaim Sheba Medical Center, Ramat Gan, Israel